CLINICAL TRIAL: NCT05531149
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center, Phase III Trial to Assess the Efficacy and Safety of Trimodulin (BT588) in Adult Hospitalized Subjects With CAP Including COVID-19 Pneumonia.
Brief Title: Efficacy and Safety of Trimodulin (BT588) in Subjects With CAP Including COVID-19 Pneumonia
Acronym: TRICOVID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unacceptable delay of trial completion Low recruitment rate
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1001
Record Dates: First submitted 2022-08-26; First posted 2022-09-07 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Infection; Pneumonia; Community-acquired Pneumonia; Acute Respiratory Distress Syndrome; COVID-19; Viral Pneumonia; Bacterial Pneumonia; Fungal Pneumonia
Keywords: Non severe community acquired pneumonia; COVID-19; SARS-CoV-2; CAP
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia; Community-Acquired Pneumonia; Respiratory Distress Syndrome; COVID-19; Pneumonia, Viral; Pneumonia, Bacterial | interventions — trimodulin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either trimodulin or placebo on a 1:1 basis, stratified by type of oxygen supply before randomization and by region
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All bottles will be indistinguishable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimodulin (Experimental): Trimodulin (human IgM, IgA, IgG solution) for intravenous (IV) administration.
  Interventions: Drug: Trimodulin
- Placebo (Placebo Comparator): Human albumin 1%
  Interventions: Drug: Placebo (human albumin 1%)

INTERVENTIONS:
Drug: Trimodulin — IMP will be administered via IV infusion on 5 consecutive days
  Other Names: BT588
  Arms: Trimodulin
Drug: Placebo (human albumin 1%) — IMP will be administered via IV infusion on 5 consecutive days
  Arms: Placebo

SUMMARY:
The main objectives of the trial are to assess the efficacy and safety of trimodulin as adjunctive treatment to standard of care (SoC) compared to placebo plus SoC in adult hospitalized subjects with non-severe community-acquired pneumonia (CAP) or moderate / severe Coronavirus Disease 2019 (COVID-19) pneumonia.

Other objectives are to determine pharmacokinetic (PK) and pharmacodynamic (PD) properties of trimodulin.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multi-center, phase III trial to assess the efficacy and safety of trimodulin compared to placebo treatment, adjunctive to SoC in adult hospitalized subjects with non-severe community-acquired pneumonia (CAP) or moderate / severe Coronavirus Disease 2019 (COVID-19) pneumonia. Patients requiring low-flow oxygen, non-invasive ventilation or high-flow oxygen and with signs of early systemic inflammation (defined by C reactive protein (CRP), D-dimer and platelet levels) will be enrolled.

Subjects will be randomized to receive either trimodulin or placebo on a 1:1 basis, stratified by type of oxygen supply before randomization and by region. Investigational Medicinal Product (IMP) treatments will be blinded. Subjects will be administered IMP once daily on five consecutive days (day 1 through day 5) adjunctive to SoC. The subsequent follow-up phase comprises maximally 23 days (day 6 through day 28) followed by an end-of-follow-up visit/telephone call on day 29 [+3]. For all subjects still in the hospital after day 29, an extended follow-up visit is conducted until day 90 or until discharge. For all subjects a closing visit/telephone call on day 91 [+10] will be done.

For the evaluation of the primary and several secondary endpoints of the trial, a 9-category ordinal scale will be used. The primary objective is to assess efficacy of trimodulin based on clinical deterioration and mortality to demonstrate superiority to treatment with placebo. Secondary objectives are to assess efficacy and safety and to determine PK and PD properties of trimodulin compared to placebo.

ELIGIBILITY:
Main Inclusion Criteria:

1. Written informed consent.
2. Hospitalized, adult (≥ 18 years of age) subjects.
3. Diagnosis of CAP or COVID- 19 pneumonia (e.g. according to local guidelines) and with radiologic evidence showing new pulmonary lobar or multilobar infiltrates consistent with CAP or COVID-19 pneumonia.
4. Receiving oxygen supply via low-flow oxygen, high-flow oxygen or on non-invasive ventilation.
5. Fulfilling at least one clinical respiratory parameter (SpO2 ≤ 94% and/or 100 mm Hg < PaO2/FiO2 ≤ 300 mm Hg).
6. Signs of early systemic inflammation based on CRP and coagulation parameter threshold levels.

Main Exclusion Criteria:

1. Pregnant or lactating women.
2. Subject on invasive mechanical ventilation and/or extracorporeal membrane oxygenation.
3. Subject with septic shock and in need for vasopressors.
4. Severe neutropenia prior to start of treatment.
5. Hemoglobin >7 g/dL prior to start of treatment.
6. Pre-existing hemolytic disease.
7. Pre-existing thromboembolic events (TEEs).
8. Subject on dialysis or with severe renal impairment prior to start of treatment.
9. Subject with end stage renal disease, or known primary focal segmental glomerulosclerosis.
10. Pre-existing severe lung diseases to current pneumonia.
11. Pre-existing decompensated heart failure.
12. Pre-existing hepatic cirrhosis, severe hepatic impairment , or hepatocellular carcinoma.
13. Known intolerance to proteins of human origin or known allergic reactions to components of trimodulin/placebo.
14. Selective, absolute immunoglobulin A (IgA) deficiency with known antibodies to IgA.
15. Known human immunodeficiency virus infection.
16. Life expectancy of less than 90 days.
17. Morbid obesity or malnutrition.
18. Treatment with predefined medications (certain immune modulators or immunosuppressants) before entering the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint | Until day 29
  Composite of percentage of subjects with a change of at least 1 category on the 9-category ordinal scale from baseline (between days 6-29) and 28-day all-cause mortality rate (between days 1-29)

SECONDARY OUTCOMES:
Clinical deterioration rate | Between days 6-29 and days 1-29
  Percentage of subjects with a change of at least 1 category on the category ordinal-scale
28-days all-cause mortality rate | Day 29
  Percentage of subjects with a change to 8 on 9-category ordinal scale.
90-days all-cause mortality rate | Day 91
  Percentage of subjects with a change to 8 on 9-category ordinal scale.
Time to recovery | Between days 1-29
  Number of days to score ≤ 2 until day 29
Proportion of subjects with score ≤ 2 | Day 29
  Proportion of subjects that improved to score ≤ 2
Proportion of subjects improved, unchanged, and deteriorated/died | Between days 1-29
  Proportion of subjects improved, unchanged, and deteriorated/died compared to baseline at several days
Proportion of subjects with different partial pressure of oxygen (PaO2)/ fraction of inspired oxygen (FiO2) ratios | Days 7, 14, 21, 29
  Proportion of subjects with PaO2/FiO2 ratio < 100, 100 to < 200, 200 to < 300 or ≥ 300
Days of invasive mechanical ventilation (IMV)/ extracorporeal membrane oxygenation (ECMO) | Day 29
  Days of IMV/ECMO
Proportion of subjects on IMV/ECMO | Day 29
  Proportion of subjects on IMV/ECMO
Days with oxygen supply | Day 29
  Days with oxygen supply
Proportion of subjects with oxygen supply | Days 7, 14, 21, 29
  Proportion of subjects with oxygen supply
Days in intensive care unit (ICU) | Day 29
  Days in intensive care unit
Proportion of subjects in ICU | Day 29
  Proportion of subjects in ICU
Days of hospitalization | Day 29
  Days of hospitalization
All adverse events (AEs), treatment-emergent AEs (TEAEs), AEs of special interest (AESIs), infusional TEAEs, TEAEs that led to permanent withdrawal of IMP and/or discontinuation of trial | Until day 29
  Number, severity, causality, outcome, and seriousness of all adverse events (AEs), treatment-emergent AEs (TEAEs), AEs of special interest (AESIs), infusional TEAEs, TEAEs that led to permanent withdrawal of IMP, and TEAEs that led to discontinuation of the trial
TEAEs | Until day 29
  Number of all related TEAEs
SAEs | Until day 29
  Number, severity, causality, and outcome of all serious adverse events (SAEs)
Dose modifications | Day 1-5
  Dose modifications (incl. reductions and changes in infusion rate)
Change over time in ECG parameters | Days -1, 1, 3, 5 and once between days 8-13
  ECG recordings, (including heart rate, QT-interval, QTcF) showing abnormal, clinically relevant findings will be reported as adverse event
Changes over time in vital signs | Days -1,1-3, 5, 7 ,14, 21, 29
  Changes in recordings of vital sign parameters showing clinically significant measurements outside the normal range will be reported as adverse event.
Changes over time in clinical laboratory parameters | Days -1, 1-5, 7,14, 21, 29
  Changes in recordings for clinical laboratory values (including chemistry, hematology and coagulation) showing clinically significant measurements outside the normal range will be reported as adverse event.

OTHER OUTCOMES:
Pharmacokinetic assessment of immunoglobulins | Day 1, 5, 14
  Assessment of changes in serum concentrations (g/L) of immunoglobulin M (IgM), immunoglobulin A (IgA), and immunoglobulin G (IgG) before, during and after treatment
Pharmacodynamic assessment of disease related serum proteins | Days 1, 3, 5, 7, 14
  Assessment of relative changes in serum concentrations from baseline before, during and after treatment including markers of inflammation, coagulation, complement factors and biomarkers (e.g. % change in Interleukin-6)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Torres, Prof, Principal Investigator — Hospital Clinic de Barcelona, Barcelona, Spain
Locations (64):
- Argentina (3):
  - Investigational Site #5401, Buenos Aires
  - Investigational Site #5403, Córdoba
  - Investigational Site #5402, Córdoba
- Austria (3):
  - Investigational Site #4303, Klagenfurt
  - Investigational Site #4302, Linz
  - Investigational Site #4304, Vienna
- Belgium (3):
  - Investigational Site #3203, Edegem
  - Investigational Site #3202, Mechelen
  - Investigational Site #3201, Ottignies
- Brazil (11):
  - Investigational Site #5508, Campo Largo, São Paulo
  - Investigational Site #5509, Ribeirão Preto, São Paulo
  - Investigational Site #5511, São Paulo, São Paulo
  - Investigational Site #5505, Botucatu
  - Investigational Site #5503, Porto Alegre
  - Investigational Site #5507, Porto Alegre
  - Investigational Site #5506, Porto Alegre
  - Investigational Site #5502, Santo André
  - Investigational Site #5510, Santos
  - Investigational Site #5504, São José do Rio Preto
  - Investigational Site #5501, São Paulo
- France (8):
  - Investigational Site #3303, Melun
  - Investigational Site #3304, Paris
  - Investigational Site #3301, Paris
  - Investigational Site #3305, Saint-Etienne
  - Investigational Site #3307, Salouël
  - Investigational Site #3306, Strasbourg
  - Investigational Site #3308, Strasbourg
  - Investigational Site #3302, Trévenans
- Germany (5):
  - Investigational Site #4904, Berlin
  - Investigational Site #4901, Bochum
  - Investogational Site #4902, Cottbus
  - Investigational Site #4903, Hanover
  - Investigational Site #4907, München
- Hungary (2):
  - Investigational SIte #3603, Debrecen
  - Investigational Site #3601, Szeged
- Latvia (2):
  - Investigational Site #7102, Daugavpils
  - Investigational Site #7101, Riga
- Lithuania (7):
  - Investigational Site #7002, Kaunas
  - Investigational Site #7007, Kaunas
  - Investigational Site #7005, Kaunas
  - Investigational Site #7003, Klaipėda
  - Investigational Site #7004, Šiauliai
  - Investigational Site #7006, Vilnius
  - Investigational Site #7001, Vilnius
- Portugal (2):
  - Investigational Site #3502, Guimarães
  - Investogational SIte #3501, Lisbon
- Slovakia (5):
  - Investigational Site #2103, Banská Bystrica
  - Investigational Site #2102, Malacky
  - Investigational Site #2105, Michalovce
  - Investigational Site #2101, Nitra
  - Investigational Site #2104, Svidník
- South Africa (7):
  - Investigational site #2706, Kimberley
  - Investigational Site #2702, Klerksdorp
  - Investigational Site #2703, Mthatha
  - Investigational Site #2705, Plettenberg Bay
  - Investigational Site #2701, Pretoria
  - Investigational Site #2707, Pretoria
  - Investigational Site #2704, Pretoria
- Spain (3):
  - Investigational Site #3401, Barcelona
  - Investigational Site #3403, Madrid
  - Investigational Site #3404, Madrona
- Turkey (Türkiye) (3):
  - Investigational Site #9005, Ankara
  - Investigational Site #9004, Istanbul
  - Investigational Site #9001, Trabzon

IPD SHARING:
Plan to Share IPD: No